CLINICAL TRIAL: NCT01702363
Title: A 52-week, Multi-centre, Open-label Study to Evaluate the Safety and Tolerability of GSK573719 125 mcg Once-daily Via Novel Dry Powder Inhaler (nDPI) in Japanese Subjects With Chronic Obstructive Pulmonary Disease.
Brief Title: Long-term Safety Study for GSK573719 in Japanese
Acronym: AC4115361
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115361
Record Dates: First submitted 2012-09-20; First posted 2012-10-08 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease (COPD), GSK573719, Pharmacogenetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK573719 (Experimental): 125mcg
  Interventions: Drug: GSK573719

INTERVENTIONS:
Drug: GSK573719 — GSK573719 inhalation powder inhaled orally once daily for 52 weeks.

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of GSK573719 Inhalation Powder 125 mcg once-daily over 52 weeks in Japanese subjects with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) treatment guidelines recommend an incremental approach to pharmacological treatment as the disease state worsens, involving the use of combinations of drug classes with different or complementary mechanisms of action [Celli, 2004, GOLD 2009]. As disease progresses from mild to moderate, regular treatment with one or more long-acting bronchodilators is recommended. Inhaled bronchodilators, including beta2 agonists and anticholinergics are included with inhaled corticosteroids (ICS) therapy and are mainstays of therapy in patients diagnosed with COPD. Since GSK573719 Inhalation Powder is expected to be used for chronic management of COPD as long-acting muscarinic antagonist (LAMA), this study is intended to evaluate the safety and tolerability of long-term administration of GSK573719 Inhalation Powder 125 mcg in Japanese patients with COPD at doses possibly used to be in Japan.

In this study, patient safety will also be monitored by evaluating pulmonary function and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient.
* A signed and dated written informed consent prior to study participation.
* Japanese subjects 40 years of age or older at Visit 1.
* Male or female subjects. A female is eligible if she is of: Non-child bearing potential or Child bearing potential agrees to one of the contraceptive methods.
* Subjects with a clinical history of COPD in accordance with the definition by COPD domestic guideline.
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Visit 1.
* Subject with a measured post-salbutamol forced expiratory volume/forced vital capacity (FEV1/FVC) ratio of <70% and Subjects with a measured post-salbutamol FEV1 <80% of predicted normal values.

Exclusion Criteria (Visit 1):

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* A current diagnosis of asthma.
* Known respiratory disorders other than COPD.
* Subjects with historical or current evidence of clinically significant abnormalities that are uncontrolled.
* A chest X-ray or computed tomography (CT) scan that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD.
* Allergy or hypersensitivity to muscarinic, beta2-agonist, lactose/milk protein or magnesium stearate or a condition that contraindicates participation.
* Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1.
* Significantly abnormal finding from clinical chemistry or hematology, tests at Visit 1.
* Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day.
* Regular use (prescribed every day, not for as-needed use) of short-acting bronchodilators (e.g., salbutamol) via nebulized therapy.
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1.
* A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site.
* Previous use of GSK573719, the GSK573719/GW642444 combination.
* Use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer).

Exclusion Criteria (Visit 2):

- COPD Exacerbation during run-in period: Subject must not have experienced a COPD exacerbation or a lower respiratory tract infection during run-in or at Visit 2.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Japan (15):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Yamagata E, Soutome T, Hashimoto K, Mihara K, Tohda Y. Long-term (52 weeks) safety and tolerability of umeclidinium in Japanese patients with chronic obstructive pulmonary disease. Curr Med Res Opin. 2016 May;32(5):967-73. doi: 10.1185/03007995.2016.1140029. Epub 2016 Feb 18. PMID 26782971
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115361 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 131 Japanese participants with chronic obstructive pulmonary disease (COPD) who met the eligibility criteria were registered and administration of investigational product was started
Pre-assignment Details: Participants entered a 7- to 14-day Run-in Period followed by a 52-week Treatment Period. Follow-up was conducted by a phone call approximately 1 week following the completion of treatment or withdrawal from the trial.
Groups:
- UMEC 125 µg QD: Participants received umeclidinium bromide (UMEC) 125 micrograms (µg) once daily (QD) in the morning via a dry powder inhaler (DPI) for 52 weeks.
Period: Overall Study
Arm/Group | UMEC 125 µg QD
Started | 131
Completed | 111
Not Completed | 20
Not completed — Adverse Event | 14
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- UMEC 125 µg QD: Participants received UMEC 125 µg QD in the morning via a DPI for 52 weeks.
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.2 (7.77)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 128
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) Throughout the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of the study medication, whether or not considered related to the study medication. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the study medication. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect, or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, or is an event of possible drug-induced liver injury. Medical or scientific judgment was exercised in deciding whether reporting was appropriate in other situations.
Time Frame: From the first dose of study medication up to 52 weeks
Population: Intent-to Treat (ITT) Population: All participants who received at least one dose of the study medication. For participants who withdrew from the study, all available data collected until the time of study discontinuation were included in the ITT analysis.
Measure: Number; unit: Participants
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Participants
  Any AE | 105
  Any SAE | 17

2. Primary Outcome: Number of Participants With AEs Classified by the Indicated Maximum Grade Severity Throughout the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of the study medication, whether or not considered related to the study medication. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the study medication. AEs were classified according to intensity based upon the investigators' clinical judgment. The intensity was categorized as: mild (an event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities); moderate (an event that is sufficiently discomforting to interfere with normal everyday activities); or severe (an event that prevents normal everyday activities).
Time Frame: From the first dose of study medication up to 52 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Participants
  Any AE, mild | 78
  Any AE, moderate | 18
  Any AE, severe | 9

3. Secondary Outcome: Basophil, Eosinophil, Lymphocyte, Monocyte, and Total Neutrophil Values at Baseline (BL) (Week -2), Week 12, Week 24, Week 36, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of the indicated laboratory parameters at the following time points: BL (Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD Visit (conducted for participants who completed the Week 24 Visit or withdrew before Week 24), and Week 52/WD Visit (conducted for participants who completed the Week 52 Visit or withdrew before Week 52). The BL value for clinical laboratory tests was the value recorded on Week -2 (Screening Visit).
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD Visit, and Week 52/WD Visit
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters and at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of cells in blood
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Percentage of cells in blood
  Basophils, BL (Week -2), n=131 | 0.62 (0.462)
  Basophils, Week 12, n=126 | 0.68 (0.494)
  Basophils, Week 24, n=121 | 0.63 (0.433)
  Basophils, Week 36, n=114 | 0.63 (0.391)
  Basophils, Week 52, n=111 | 0.64 (0.455)
  Basophils, WD Visit, n=15 | 0.61 (0.516)
  Basophils, Week 24/WD, n=128 | 0.63 (0.446)
  Basophils, Week 52/WD, n=126 | 0.63 (0.460)
  Eosinophils, BL (Week -2), n=131 | 3.74 (3.573)
  Eosinophils, Week 12, n=126 | 3.61 (2.451)
  Eosinophils, Week 24, n=121 | 3.74 (3.453)
  Eosinophils, Week 36, n=114 | 3.69 (2.903)
  Eosinophils, Week 52, n=111 | 3.93 (4.188)
  Eosinophils, WD Visit, n=15 | 2.94 (3.715)
  Eosinophils, Week 24/WD, n=128 | 3.61 (3.424)
  Eosinophils, Week 52/WD, n=126 | 3.81 (4.133)
  Lymphocytes, BL (Week -2), n=131 | 30.96 (7.711)
  Lymphocytes, Week 12, n=126 | 29.53 (7.340)
  Lymphocytes, Week 24, n=121 | 29.98 (7.214)
  Lymphocytes, Week 36, n=114 | 30.76 (6.840)
  Lymphocytes, Week 52, n=111 | 29.87 (6.622)
  Lymphocytes, WD Visit, n=15 | 23.58 (10.609)
  Lymphocytes, Week 24/WD, n=128 | 29.26 (8.001)
  Lymphocytes, Week 52/WD, n=126 | 29.12 (7.442)
  Monocytes, BL (Week -2), n=131 | 6.35 (1.494)
  Monocytes, Week 12, n=126 | 6.25 (1.516)
  Monocytes, Week 24, n=121 | 6.39 (1.751)
  Monocytes, Week 36, n=114 | 6.25 (1.539)
  Monocytes, Week 52, n=111 | 6.45 (1.727)
  Monocytes, WD Visit, n=15 | 5.83 (2.264)
  Monocytes, Week 24/WD, n=128 | 6.34 (1.848)
  Monocytes, Week 52/WD, n=126 | 6.38 (1.800)
  Total Neutrophils, BL (Week -2), n=131 | 58.34 (7.818)
  Total Neutrophils, Week 12, n=126 | 59.93 (8.065)
  Total Neutrophils, Week 24, n=121 | 59.26 (8.273)
  Total Neutrophils, Week 36, n=114 | 58.67 (7.219)
  Total Neutrophils, Week 52, n=111 | 59.11 (7.107)
  Total Neutrophils, WD Visit, n=15 | 67.04 (14.099)
  Total Neutrophils, Week 24/WD, n=128 | 60.16 (9.378)
  Total Neutrophils, Week 52/WD, n=126 | 60.05 (8.565)

4. Secondary Outcome: Eosinophil Values, Total Neutrophil Values, Platelet Count, and White Blood Cell (WBC) Count at BL (Week -2), Week 12, Week 24, Week 36, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of the indicated laboratory parameters at the following time points: BL (Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 Visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 Visit or withdrew before Week 52). The BL value for clinical laboratory tests was the value recorded on Week -2 (Screening Visit).
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter (GI/L)
Groups:
- MEC 125 µg QD: Participants received UMEC 125 µg QD in the morning via a DPI for 52 weeks.
Arm/Group | MEC 125 µg QD
Number analyzed (Participants) | 131
10^9 cells per Liter (GI/L)
  Eosinophils, BL (Week -2), n=131 | 0.222 (0.1808)
  Eosinophils, Week 12, n=126 | 0.213 (0.1426)
  Eosinophils, Week 24, n=121 | 0.218 (0.1958)
  Eosinophils, Week 36, n=114 | 0.215 (0.1542)
  Eosinophils, Week 52, n=111 | 0.233 (0.2074)
  Eosinophils, WD Visit, n=15 | 0.189 (0.2265)
  Eosinophils, Week 24/WD, n=128 | 0.210 (0.1947)
  Eosinophils, Week 52/WD, n=126 | 0.228 (0.2093)
  Total Neutrophils, BL (Week -2), n=131 | 3.673 (1.1732)
  Total Neutrophils, Week 12, n=126 | 3.705 (1.1894)
  Total Neutrophils, Week 24, n=121 | 3.639 (1.2147)
  Total Neutrophils, Week 36, n=114 | 3.576 (1.1978)
  Total Neutrophils, Week 52, n=111 | 3.709 (1.1155)
  Total Neutrophils, WD Visit, n=15 | 4.657 (2.3277)
  Total Neutrophils, Week 24/WD, n=128 | 3.709 (1.4098)
  Total Neutrophils, Week 52/WD, n=126 | 3.821 (1.3405)
  Platelet Count, BL (Week -2), n=131 | 228.8 (55.42)
  Platelet Count, Week 12, n=126 | 232.1 (57.03)
  Platelet Count, Week 24, n=121 | 228.3 (53.74)
  Platelet Count, Week 36, n=114 | 224.6 (51.22)
  Platelet Count, Week 52, n=111 | 229.3 (52.38)
  Platelet Count, WD Visit, n=15 | 217.3 (48.02)
  Platelet Count, Week 24/WD, n=128 | 226.9 (54.03)
  Platelet Count, Week 52/WD, n=126 | 227.9 (51.85)
  WBC Count, BL (Week -2), n=131 | 6.24 (1.594)
  WBC Count, Week 12, n=126 | 6.13 (1.549)
  WBC Count, Week 24, n=121 | 6.07 (1.544)
  WBC Count, Week 36, n=114 | 6.04 (1.552)
  WBC Count, Week 52, n=111 | 6.23 (1.558)
  WBC Count, WD Visit, n=15 | 6.87 (2.456)
  WBC Count, Week 24/WD, n=128 | 6.08 (1.664)
  WBC Count, Week 52/WD, n=126 | 6.31 (1.690)

5. Secondary Outcome: Hemoglobin, Albumin, and Total Protein Values at BL (Week -2), Week 12, Week 24, Week 36, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: as for outcome 4
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Grams per Liter (G/L)
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Grams per Liter (G/L)
  Hemoglobin, BL (Week -2), n=131 | 146.2 (13.66)
  Hemoglobin, Week 12, n=126 | 147.4 (13.96)
  Hemoglobin, Week 24, n=121 | 147.3 (13.59)
  Hemoglobin, Week 36, n=114 | 145.6 (12.39)
  Hemoglobin, Week 52, n=111 | 147.8 (13.39)
  Hemoblobin, WD Visit, n=15 | 134.4 (13.92)
  Hemoglobin, Week 24/WD, n=128 | 146.5 (14.19)
  Hemoglobin, Week 52/WD, n=126 | 146.2 (14.09)
  Albumin, BL (Week -2), n=131 | 41.9 (2.91)
  Albumin, Week 12, n=126 | 42.5 (3.06)
  Albumin, Week 24, n=121 | 42.3 (3.05)
  Albumin, Week 36, n=114 | 42.3 (2.94)
  Albumin, Week 52, n=111 | 42.6 (3.06)
  Albumin, WD Visit, n=15 | 38.9 (3.13)
  Albumin, Week 24/WD, n=128 | 42.1 (3.18)
  Albumin, Week 52/WD, n=126 | 42.2 (3.29)
  Total Protein, BL (Week -2), n=131 | 70.4 (4.05)
  Total Protein, Week 12, n=126 | 70.9 (4.13)
  Total Protein, Week 24, n=121 | 70.8 (4.09)
  Total Protein, Week 36, n=114 | 70.0 (4.36)
  Total Protein, Week 52, n=111 | 70.4 (4.42)
  Total Protein, WD Visit, n=15 | 67.7 (4.67)
  Total Protein, Week 24/WD, n=128 | 70.6 (4.23)
  Total Protein, Week 52/WD, n=126 | 70.1 (4.52)

6. Secondary Outcome: Hematocrit Values at BL (Week -2), Week 12, Week 24, Week 36, Week 52, the Withdrawal (WD) Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of hematocrit at the following time points: BL (Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 Visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 Visit or withdrew before Week 52). The BL value for clinical laboratory tests was the value recorded on Week -2 (Screening Visit).
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Proportion of red blood cells in blood
  BL (Week -2), n=131 | 0.4457 (0.03961)
  Week 12, n=126 | 0.4511 (0.04075)
  Week 24, n=121 | 0.4513 (0.03895)
  Week 36, n=114 | 0.4434 (0.03628)
  Week 52, n=111 | 0.4419 (0.03726)
  WD Visit, n=15 | 0.4124 (0.04371)
  Week 24/WD, n=128 | 0.4484 (0.04108)
  Week 52/WD, n=126 | 0.4384 (0.03909)

7. Secondary Outcome: Alkaline Phosphatase (AP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Creatine Kinase, and Gamma Glutamyl Transferase (GGT) Values at BL (Week -2), Week 12, Week 24, Week 36, Week 52, the WD Visit, Week 24/WD, and Week 52/WD
Description: as for outcome 4
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
International Units per Liter (IU/L)
  AP, BL (Week -2), n=131 | 233.1 (61.19)
  AP, Week 12, n=126 | 239.2 (68.51)
  AP, Week 24, n=121 | 237.5 (63.33)
  AP, Week 36, n=114 | 232.4 (65.73)
  AP, Week 52, n=111 | 235.1 (64.83)
  AP, WD Visit, n=15 | 258.0 (83.49)
  AP, Week 24/WD, n=128 | 239.4 (67.27)
  AP, Week 52/WD, n=126 | 237.8 (67.34)
  ALT, BL (Week -2), n=131 | 21.1 (11.25)
  ALT, Week 12, n=126 | 20.2 (9.70)
  ALT, Week 24, n=121 | 19.9 (10.45)
  ALT, Week 36, n=114 | 20.1 (11.94)
  ALT, Week 52, n=111 | 20.7 (10.34)
  ALT, WD Visit, n=15 | 23.9 (27.36)
  ALT, Week 24/WD, n=128 | 20.5 (13.62)
  ALT, Week 52/WD, n=126 | 21.1 (13.38)
  AST, BL (Week -2), n=131 | 23.7 (11.72)
  AST, Week 12, n=126 | 23.0 (8.46)
  AST, Week 24, n=121 | 22.2 (7.12)
  AST, Week 36, n=114 | 22.5 (11.72)
  AST, Week 52, n=111 | 23.2 (8.10)
  AST, WD Visit, n=15 | 28.7 (25.04)
  AST, Week 24/WD, n=128 | 23.1 (10.97)
  AST, Week 52/WD, n=126 | 23.8 (11.45)
  Creatine Kinase, BL (Week -2), n=131 | 124.8 (71.56)
  Creatine Kinase, Week 12, n=126 | 119.7 (92.39)
  Creatine Kinase, Week 24, n=121 | 117.3 (70.74)
  Creatine Kinase, Week 36, n=114 | 113.8 (70.26)
  Creatine Kinase, Week 52, n=111 | 109.5 (60.10)
  Creatine Kinase, WD Visit, n=15 | 144.7 (147.28)
  Creatine Kinase, Week 24/WD, n=128 | 119.8 (82.66)
  Creatine Kinase, Week 52/WD, n=126 | 113.7 (75.76)
  GGT, BL (Week -2), n=131 | 40.1 (38.68)
  GGT, Week 12, n=126 | 38.1 (34.09)
  GGT, Week 24, n=121 | 39.5 (42.83)
  GGT, Week 36, n=114 | 40.0 (44.18)
  GGT, Week 52, n=111 | 42.2 (49.47)
  GGT, WD Visit, n=15 | 49.5 (77.05)
  GGT, Week 24/WD, n=128 | 40.9 (48.86)
  GGT, Week 52/WD, n=126 | 43.1 (53.14)

8. Secondary Outcome: Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Creatinine, and Uric Acid Values at BL (Week -2), Week 12, Week 24, Week 36, Week 52, the WD Visit, Week 24/WD, and Week 52/WD
Description: as for outcome 4
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (µM/L)
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Micromoles per Liter (µM/L)
  Direct Bilirubin, BL (Week -2), n=131 | 3.577 (2.0172)
  Direct Bilirubin, Week 12, n=126 | 3.284 (1.6699)
  Direct Bilirubin, Week 24, n=121 | 3.137 (1.5508)
  Direct Bilirubin, Week 36, n=114 | 3.450 (1.7323)
  Direct Bilirubin, Week 52, n=111 | 3.389 (1.6783)
  Direct Bilirubin, WD Visit, n=15 | 3.192 (1.4258)
  Direct Bilirubin, Week 24/WD, n=128 | 3.153 (1.5539)
  Direct Bilirubin, Week 52/WD, n=126 | 3.366 (1.6464)
  Indirect Bilirubin, BL (Week -2), n=131 | 6.305 (2.8933)
  Indirect Bilirubin, Week 12, n=126 | 6.664 (2.8271)
  Indirect Bilirubin, Week 24, n=121 | 6.444 (2.8077)
  Indirect Bilirubin, Week 36, n=114 | 6.975 (3.4662)
  Indirect Bilirubin, Week 52, n=111 | 6.948 (3.0176)
  Indirect Bilirubin, WD Visit, n=15 | 5.814 (3.0861)
  Indirect Bilirubin, Week 24/WD, n=128 | 6.426 (2.8930)
  Indirect Bilirubin, Week 52/WD, n=126 | 6.813 (3.0358)
  Total Bilirubin, BL (Week -2), n=131 | 9.881 (4.4353)
  Total Bilirubin, Week 12, n=126 | 9.948 (4.0720)
  Total Bilirubin, Week 24, n=121 | 9.582 (3.9273)
  Total Bilirubin, Week 36, n=114 | 10.425 (4.7718)
  Total Bilirubin, Week 52, n=111 | 10.337 (4.3954)
  Total Bilirubin, WD Visit, n=15 | 9.006 (4.3099)
  Total Bilirubin, Week 24/WD, n=128 | 9.579 (4.0337)
  Total Bilirubin, Week 52/WD, n=126 | 10.179 (4.3896)
  Creatinine, BL (Week -2), n=131 | 73.1088 (15.62560)
  Creatinine, Week 12, n=126 | 73.5965 (16.73127)
  Creatinine, Week 24, n=121 | 73.1894 (15.82538)
  Creatinine, Week 36, n=114 | 73.2092 (15.29351)
  Creatinine, Week 52, n=111 | 72.3287 (14.54036)
  Creatinine, WD Visit, n=15 | 78.0277 (26.02168)
  Creatinine, Week 24/WD, n=128 | 73.3789 (16.14369)
  Creatinine, Week 52/WD, n=126 | 73.0072 (16.28875)
  Uric Acid, BL (Week -2), n=131 | 347.9353 (81.78271)
  Uric Acid, Week 12, n=126 | 336.5813 (78.06630)
  Uric Acid, Week 24, n=121 | 346.9011 (78.45280)
  Uric Acid, Week 36, n=114 | 352.6016 (81.62589)
  Uric Acid, Week 52, n=111 | 343.4836 (67.79140)
  Uric Acid, WD Visit, n=15 | 343.3979 (96.73417)
  Uric Acid, Week 24/WD, n=128 | 344.4264 (78.41134)
  Uric Acid, Week 52/WD, n=126 | 343.4734 (71.35989)

9. Secondary Outcome: Calcium, Chloride, Glucose, Carbon Dioxide/Bicarbonate (CO2/HCO3), Potassium, Sodium, Inorganic Phosphorus, and Urea/Blood Urea Nitrogen (Urea/BUN) Values at BL (Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Description: Blood samples were collected for the measurement of the indicated laboratory parameters at the following time points: BL (Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit (conducted for participants who withdrew at any point during the study), Week 24/WD (conducted for participants who completed the Week 24 Visit or withdrew before Week 24), and Week 52/WD (conducted for participants who completed the Week 52 Visit or withdrew before Week 52). The Baseline value for clinical laboratory tests was the value recorded on Week -2 (Screening Visit).
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD, and Week 52/WD
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (MMOL/L)
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Millimoles per Liter (MMOL/L)
  Calcium, BL (Week -2), n=131 | 2.2804 (0.09567)
  Calcium, Week 12, n=126 | 2.2720 (0.09628)
  Calcium, Week 24, n=121 | 2.2589 (0.10287)
  Calcium, Week 36, n=114 | 2.2505 (0.09407)
  Calcium, Week 52, n=111 | 2.2680 (0.09580)
  Calcium, WD Visit, n=15 | 2.1923 (0.09281)
  Calcium, Week 24/WD, n=128 | 2.2556 (0.10334)
  Calcium, Week 52/WD, n=126 | 2.2590 (0.09822)
  Chloride, BL (Week -2), n=131 | 103.2 (2.58)
  Chloride, Week 12, n=126 | 103.0 (2.61)
  Chloride, Week 24, n=121 | 103.0 (2.89)
  Chloride, Week 36, n=114 | 104.2 (3.26)
  Chloride, Week 52, n=111 | 104.1 (2.74)
  Chloride, WD Visit, n=15 | 104.1 (4.61)
  Chloride, Week 24/WD, n=128 | 103.0 (3.06)
  Chloride, Week 52/WD, n=126 | 104.1 (2.99)
  Glucose, BL (Week -2), n=131 | 5.9980 (1.55438)
  Glucose, Week 12, n=126 | 6.3127 (1.91203)
  Glucose, Week 24, n=121 | 6.2735 (1.75968)
  Glucose, Week 36, n=114 | 6.6047 (2.23873)
  Glucose, Week 52, n=111 | 6.3957 (1.88553)
  Glucose, WD Visit, n=15 | 6.9721 (2.28881)
  Glucose, Week 24/WD, n=128 | 6.3364 (1.83801)
  Glucose, Week 52/WD, n=126 | 6.4643 (1.93661)
  CO2/HCO3, BL (Week -2), n=131 | 24.7 (1.95)
  CO2/HCO3, Week 12, n=126 | 24.2 (1.85)
  CO2/HCO3, Week 24, n=121 | 24.0 (2.17)
  CO2/HCO3, Week 36, n=114 | 22.6 (2.18)
  CO2/HCO3, Week 52, n=111 | 22.8 (2.16)
  CO2/HCO3, WD Visit, n=15 | 22.9 (2.09)
  CO2/HCO3, Week 24/WD, n=128 | 24.0 (2.14)
  CO2/HCO3, Week 52/WD, n=126 | 22.8 (2.14)
  Potassium, BL (Week -2), n=131 | 4.28 (0.322)
  Potassium, Week 12, n=126 | 4.34 (0.309)
  Potassium, Week 24, n=121 | 4.32 (0.359)
  Potassium, Week 36, n=114 | 4.26 (0.345)
  Potassium, Week 52, n=111 | 4.23 (0.325)
  Potassium, WD Visit, n=15 | 4.21 (0.261)
  Potassium, Week 24/WD, n=128 | 4.31 (0.355)
  Potassium, Week 52/WD, n=126 | 4.23 (0.317)
  Sodium, BL (Week -2), n=131 | 141.5 (1.99)
  Sodium, Week 12, n=126 | 141.6 (1.97)
  Sodium, Week 24, n=121 | 142.0 (1.98)
  Sodium, Week 36, n=114 | 141.6 (1.90)
  Sodium, Week 52, n=111 | 141.0 (1.95)
  Sodium, WD Visit, n=15 | 140.8 (2.98)
  Sodium, Week 24/WD, n=128 | 141.9 (2.17)
  Sodium, Week 52/WD, n=126 | 141.0 (2.09)
  Inorganic Phosphorus , BL (Week -2), n=131 | 0.9707 (0.14747)
  Inorganic Phosphorus, Week 12, n=126 | 0.9731 (0.14204)
  Inorganic Phosphorus, Week 24, n=121 | 0.9895 (0.14258)
  Inorganic Phosphorus, Week 36, n=114 | 0.9942 (0.14571)
  Inorganic Phosphorus, Week 52, n=111 | 0.9888 (0.15944)
  Inorganic Phosphorus, WD Visit, n=15 | 0.9687 (0.18388)
  Inorganic Phosphorus, Week 24/WD, n=128 | 0.9853 (0.14531)
  Inorganic Phosphorus, Week 52/WD, n=126 | 0.9864 (0.16187)
  Urea/BUN, BL (Week -2), n=131 | 5.2945 (1.72055)
  Urea/BUN, Week 12, n=126 | 5.4556 (1.50863)
  Urea/BUN, Week 24, n=121 | 5.4072 (1.44057)
  Urea/BUN, Week 36, n=114 | 5.4386 (1.73080)
  Urea/BUN, Week 52, n=111 | 5.1788 (1.37133)
  Urea/BUN, WD Visit, n=15 | 6.2546 (2.28218)
  Urea/BUN, Week 24/WD, n=128 | 5.4551 (1.48499)
  Urea/BUN, Week 52/WD, n=126 | 5.3068 (1.53642)

10. Secondary Outcome: Change From BL in Blood Pressure Throughout the Treatment Period
Description: Blood pressure measurements included systolic blood pressure (SBP) and diastolic blood pressure (DBP). Blood pressure was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Change from BL was calculated as the assessment value at the time of interest minus the BL value. The BL value was recorded at Week 0. The WD Visit was conducted for participants who withdrew at any point during the study. The Week 24/WD Visit was conducted for participants who completed the Week 24 Visit or withdrew before Week 24. The Week 52/WD Visit was conducted for participants who completed the Week 52 Visit or withdrew before Week 52.
Time Frame: BL(Week 0), Week 4, Week 8, Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD Visit, and Week 52/WD Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
millimeters of mercury (mmHg)
  SBP, Week 4, n=128 | 2.2 (12.47)
  SBP, Week 8, n=127 | 4.1 (13.06)
  SBP, Week 12, n=126 | 3.3 (15.14)
  SBP, Week 24, n=121 | 2.6 (15.18)
  SBP, Week 36, n=114 | -1.1 (16.78)
  SBP, Week 52, n=111 | -0.5 (14.95)
  SBP, WD Visit, n=17 | -2.4 (20.96)
  SBP, Week 24/WD, n=129 | 2.0 (16.19)
  SBP, Week 52/WD, n=128 | -0.8 (15.79)
  DBP, Week 4, n=128 | 0.4 (9.98)
  DBP, Week 8, n=127 | 1.6 (10.40)
  DBP, Week 12, n=126 | 1.2 (10.63)
  DBP, Week 24, n=121 | 1.3 (9.86)
  DBP, Week 36, n=114 | -1.3 (11.24)
  DBP, Week 52, n=111 | -1.3 (9.29)
  DBP, WD Visit, n=17 | -0.4 (11.50)
  DBP, Week 24/WD, n=129 | 0.9 (10.15)
  DBP, Week 52/WD, n=128 | -1.2 (9.57)

11. Secondary Outcome: Change From BL in Heart Rate Throughout the Treatment Period
Description: Heart rate was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Change from BL was calculated as the assessment value at the time of interest minus the BL value. The BL value was recorded at Week 0. The WD Visit was conducted for participants who withdrew at any point during the study. The Week 24/WD Visit was conducted for participants who completed the Week 24 Visit or withdrew before Week 24. The Week 52/WD Visit was conducted for participants who completed the Week 52 Visit or withdrew before Week 52.
Time Frame: BL (Week 0), Week 4, Week 8, Week 12, Week 24, Week 36, Week 52, WD Visit, Week 24/WD Visit, and Week 52/WD Visit
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters or at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
beats per minute
  Week 4, n=128 | 0.1 (9.36)
  Week 8, n=127 | -0.3 (11.07)
  Week 12, n=126 | -1.4 (9.71)
  Week 24, n=121 | -0.1 (9.42)
  Week 36, n=114 | -1.8 (10.84)
  Week 52, n=111 | -0.4 (9.72)
  WD Visit, n=17 | 7.8 (30.78)
  Week 24/WD, n=129 | 1.0 (14.17)
  Week 52/WD, n=128 | 0.7 (14.46)

12. Secondary Outcome: Number of Participants With Abnormal Findings in 12-lead Electrocardiograms (ECG) at the Indicated Time Points
Description: A 12-lead ECG was recorded in a supine position after the participant was kept at rest in this position for at least 5 minutes. Data are presented as clinically significant (CS) or not clinically significant (NCS) abnormal findings. An abnormal and significant ECG finding includes the presence of a QT interval corrected for heart rate (QTc interval) >500 milliseconds (msec) or an uncorrected QT interval >600 msec, for participants with Bundle Branch Block QTc >530 msec based on an average QTc value of triplicate ECGs. The study investigator determined if the abnormal ECG finding was CS or NCS. The WD Visit was conducted for participants who withdrew at any point during the study. The Week 24/WD and Week 52/WD Visits were conducted for participants who completed the Week 24 Visit or withdrew before Week 24 and completed the Week 52 Visit or withdrew before Week 52, respectively. The BL value for clinical laboratory tests was the value recorded on Week -2 (Screening Visit).
Time Frame: BL (Screening Visit: Week -2), Week 12, Week 24,Week 36, Week 52, WD Visit, Week 24/WD Visit, and Week 52/WD Visit
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Number; unit: Participants
Arm/Group | UMEC 125 µg QD
Number analyzed (Participants) | 131
Participants
  BL (Week -2) Abnormal NCS, n=131 | 57
  BL (Week -2), Abnormal CS, n=131 | 1
  Week 12, Abnormal NCS, n=126 | 55
  Week 12, Abnormal CS, n=126 | 0
  Week 24, Abnormal NCS, n=121 | 50
  Week 24, Abnormal CS, n=121 | 0
  Week 36, Abnormal NCS, n=114 | 45
  Week 36, Abnormal CS, n=114 | 0
  Week 52, Abnormal NCS, n=111 | 50
  Week 52, Abnormal CS, n=111 | 0
  WD Visit, Abnormal NCS, n=16 | 8
  WD Visit, Abnormal CS, n=16 | 1
  Week 24/WD, Abnormal NCS, n=128 | 53
  Week 24/WD, Abnormal CS, n=128 | 1
  Week 52/WD, Abnormal NCS, n=127 | 58
  Week 52/WD, Abnormal CS, n=127 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up (up to 53 weeks).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants who had received one dose of study drug.
Arm/Group | UMEC 125 µg QD
Serious Adverse Events (participants affected / at risk) | 17/131
Other Adverse Events (participants affected / at risk) | 71/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 125 µg QD (N=131)
Pneumonia (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Cerebellar haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Hypothermia (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Fractured ischium (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 125 µg QD (N=131)
Nasopharyngitis (Infections and infestations) | 42
Bronchitis (Infections and infestations) | 10
Pharyngitis (Infections and infestations) | 9
Pneumonia (Infections and infestations) | 9
Constipation (Gastrointestinal disorders) | 11
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.